CLINICAL TRIAL: NCT06035055
Title: The Feasibility of Ceftolozane/Tazobactam Continuous Infusion for Exacerbations of Cystic Fibrosis and Bronchiectasis Treated in an Outpatient Parenteral Antibiotic Therapy (OPAT) Setting
Brief Title: Ceftolozane/Tazobactam Continuous Infusion for Infective Exacerbations of Cystic Fibrosis and Bronchiectasis
Acronym: CERTAIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Coast Hospital and Health Service (Other)
Collaborators: The Prince Charles Hospital (Other Government); Mater (Other)
Responsible Party: Principal Investigator, Julia Bashford, Dr, Sunshine Coast Hospital and Health Service
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1295-4030; CT-2023-CTN-00033-1-v1 (Other: Therapeutic Goods Administration (Australia))
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Bronchiectasis; Cystic Fibrosis; Pseudomonas Aeruginosa; Burkholderia Cepacia Infection
MeSH Terms: conditions — Bronchiectasis; Cystic Fibrosis; Pseudomonas Infections; Burkholderia Infections | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Intervention Model Description: 30 patients will be recruited and will receive the study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ceftolozane/tazobactam 9g infusion (Experimental): 9g ceftolozane/tazobactam in 240 millilitres 0.9% sodium chloride IV infusion given over 24 hours for 10-14 days
  Interventions: Drug: Ceftolozane/tazobactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — 9g ceftolozane/tazobactam in 240 millilitres 0.9% sodium chloride IV infusion given over 24 hours for 10-14 days

SUMMARY:
The goal of this clinical trial is to assess the feasibility of ceftolozane/tazobactam (C/T) administered on an outpatient parenteral antibiotic therapy programme to patients with a current infective exacerbation of bronchiectasis or cystic fibrosis related to pseudomonas aeruginosa or burkholderia cepacia spp. organisms. The main question[s] it aims to answer are:

* Is C/T effective, safe, well-tolerated and able to induce clinical and microbiologic response?
* What are mechanisms of antimicrobial resistance are induced by administration of C/T?

DETAILED DESCRIPTION:
For patients with cystic fibrosis (CF) and non-CF bronchiectasis, chronic airway infection with Gram-negative organisms such as Pseudomonas aeruginosa and Burkholderia cepacia complex species (BCC) is highly challenging to treat and associated with significant morbidity and mortality. These organisms are naturally resistant towards many antibiotic classes, limiting the available arsenal of effective antibiotics for their treatment and eradication. Therefore, there is a pressing need for new antimicrobial therapy options for infective exacerbations associated with these organisms.

There are clear logistical and financial benefits for acute infective exacerbations of CF and non-CF bronchiectasis to be managed on OPAT programs. Many acute infective exacerbations can be safely managed in this way, and a substantial body of evidence supports non-inferiority of OPAT compared with inpatient care. From a logistical perspective, feasibility of OPAT programs is greatly improved by antibiotics being infused over a 24-hour period rather than via bolus several times per day. Unfortunately, many mainstay anti-pseudomonal and anti-Burkholderia antibiotics (including meropenem, imipenem and ceftazidime) are not stable for 24 hours at room/body temperature therefore are unsuitable for use on OPAT.

This study aims to assess viability of ceftolozane/tazobactam (C/T) administered via OPAT in adult patients with exacerbations of CF or non-CF bronchiectasis. Secondary aims are to describe clinical outcomes of patients receiving C/T, tolerability of C/T, relative sputum bacterial load throughout treatment and assess development of resistance to C/T and other antibiotics. We aim to recruit 30 patients, colonized with either pseudomonas aeruginosa or burkholderia cepacia complex, with a current infectious exacerbation requiring intravenous antibiotic treatment. We propose to administer C/T via infusion for 10-14 days with review at day 0-3, 5-7 and 10-14. Blood testing, sputum testing, lung function testing, administration of CF- and bronchiectasis-specific questionnaires and adverse event reporting will be carried out at these times. Serum levels of C/T will be monitored using a validated assay. Clinical review at day 28-42 will be carried out to assess for recrudescence of symptoms and further need for antibiotics and a follow-up phone call will be made at 3 months to assess whether any further antibiotics were needed for new/recrudescent symptoms of infection.

We expect to find that C/T is safe, well-tolerated and effective in treating infective exacerbations of bronchiectasis in OPAT settings. We expect to find that bacterial density in sputum samples reduces over the course of treatment, and that development of antimicrobial resistance is minimal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF or non-CF bronchiectasis
* Colonised with P. aeruginosa or BCC species
* Current infectious exacerbation requiring treatment with intravenous antibiotics
* Productive of sputum

Exclusion Criteria:

* Unable to consent
* Active pregnancy (as confirmed by urine beta-HCG)
* Not appropriate for OPAT (as determined by treating clinician)
* Estimated Creatinine Clearance < 50 millilitres/min
* History of hypersensitivity reaction to piperacillin/tazobactam or members of the cephalosporin class of antibiotics
* Unable to expectorate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the use of ceftolozane/tazobactam given via continuous infusion in an OPAT setting for the treatment of acute exacerbations of CF and bronchiectasis. | Day 0 to day 90 post commencement of intervention.
  The feasibility of the use of ceftolozane/tazobactam given via continuous infusion in an OPAT setting for the treatment of acute exacerbations of CF and bronchiectasis will be assessed. Feasibility will be determined as a composite of clinical response (as assessed by disease-specific questionnaires, serum inflammatory marker monitoring and spirometry in the case of patients with cystic fibrosis), adverse events and report of relapse of respiratory infection at 3 months.

SECONDARY OUTCOMES:
Safety and tolerability | Day 0 to day 90 post commencement of intervention.
  Safety and tolerability of continuous infusion ceftolozane/tazobactam. Ceftolozane/tazobactam has a very similar adverse event (AE) profile to other broad spectrum intravenous antibiotics, e.g. piperacillin/tazobactam and meropenem. Possible symptomatic AE's include: nausea, diarrhoea, headache, vomiting, constipation, insomnia, rash and fever. These will be assessed direct questioning of participants at the time of research visits, by clinical examination and and by participants self-reporting symptoms of concern to the research team any time during or after their course of ceftolozane/tazobactam. Possible laboratory abnormalities include: liver function test derangement and acute kidney injury. These will be monitored by regular blood tests during and after the course of ceftolozane/tazobactam.
Relative bacterial load | Day 0-1, Day 5-7, Day 10-14, Day 28-42
  To describe relative bacterial load over the course of ceftolozane/tazobactam treatment as assessed by quantitative PCR (qPCR) on sputa.
In vitro antimicrobial susceptibility/resistance | Day 0-1, Day 5-7, Day 10-14, Day 28-42
  To describe in vitro antimicrobial susceptibility of airway pathogens to ceftolozane/tazobactam and other anti-pseudomonal/anti-Burkholderia antibiotics over the course of ceftolozane/tazobactam treatment. This will be determined by a composite outcome of antimicrobial susceptibility testing, whole-genome sequencing (WGS), culturomic sequencing, and bioinformatic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Julia J Bashford, BSc, MBBS, Principal Investigator — Sunshine Coast University Hospital; Andrew Burke, MBBS, Principal Investigator — The Prince Charles Hospital

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified, line-by-line data will be be provided to researchers who provide a sound proposal to allow for meta-analyses requiring individual participant data (IPD). Data will be available immediately following publication, with there being no pre-determined end date on IPD sharing.
Time Frame: Data will be available immediately following publication, with there being no pre-determined end date on IPD sharing.
Access Criteria: Data will be available only to researchers who provide a sound proposal e.g. planned systematic review and meta-analysis.